CLINICAL TRIAL: NCT00818649
Title: Phase II Trial of Velcade Plus Vorinostat in the Treatment of High Risk MDS and Relapsed/Refractory AML
Brief Title: Bortezomib and Vorinostat in Treating Patients With High-Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met protocol stop rule [i.e., extreme toxicity]
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS044; MT2008-06R (Other: Blood and Marrow Transplantation Program); 0808M44081 (Other: IRB, University of Minnesota); MILLENNIUM-X05269 (Other: Millennium Pharmaceuticals, Inc.)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia with excess blasts; adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute minimally differentiated myeloid leukemia (M0); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities | interventions — Bortezomib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade + Vorinostat (Experimental): This is a phase II two stage single arm study combining Velcade on days 1, 4, 8, and 11 plus oral Vorinostat days 1-14 of a 21 days cycle. Treatment will continue for a total of 3 treatment cycles.
  Interventions: Drug: bortezomib; Drug: vorinostat

INTERVENTIONS:
Drug: bortezomib — 1.3mg/m^2 via peripheral subcutaneous administration on day 1, 4, 8, 11 of a 21 day cycle
  Other Names: Velcade
Drug: vorinostat — 400 mg orally (po) every day on days 1-14 of a 21 day cycle
  Other Names: suberoylanilide hydroxamic acid (SAHA)

SUMMARY:
RATIONALE: Bortezomib and vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bortezomib together with vorinostat may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with vorinostat works in treating patients with high-risk myelodysplastic syndrome or acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the clinical response to bortezomib and vorinostat in patients with high-risk myelodysplastic syndromes or acute myeloid leukemia, as defined by the International Working Group response criteria.

Secondary

* To characterize the quantitative and qualitative toxicities of this regimen in these patients.
* To assess the effect of this regimen on natural killer (NK) cell function, in terms of activating and inhibitory receptor alterations, target cell ligand and HLA class I modulation, and NK-mediated cell killing.
* To correlate the above changes with clinical response.

OUTLINE: Patients receive bortezomib subcutaneously (SQ) on days 1, 4, 8, and 11 and oral vorinostat once daily on days 1-14. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response, partial response, or hematologic improvement may receive 3 additional courses of therapy (for a maximum of 6 courses).

Bone marrow and peripheral blood samples are collected at baseline and at the completion of 3 courses of therapy for analysis of target cells (myeloid blasts) (i.e., HLA class I receptor analysis and natural killer [NK] cell receptor ligand analysis) and analysis of activating NK cell receptor alterations and NK-mediated cell killing.

After completion of study treatment, patients are followed periodically for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

Disease Specific Criteria: Pathologic Diagnosis must be confirmed by University of Minnesota Hematopathology

* Myelodysplastic Syndrome (MDS): By IPSS Category: INT-2 or High risk, By WHO Classification: RAEB-1 or RAEB-2,By cytogenetics: High Risk Cytogenetic Abnormality Present as defined by the presence Monosomy 7 or complex karyotype. Patients will be eligible after progressing through standard therapy with either Azacitidine or Decitabine. Patients with a history of 5q minus syndrome may be eligible after progressing through treatment with Lenalidomide.
* Acute Myelogenous Leukemia (AML): Histologic subtypes M0,M1,M2,M4,M5,M6,M7 are eligible and must meet one of the three criteria below:

  * Refractory Disease/Induction Failure: Failure to achieve initial remission after 2 lines of induction therapy.
  * Relapsed Disease
  * Newly diagnosed/untreated AML: Patients who are not able to tolerate potentially curative conventional induction chemotherapy due to advanced age, end organ limitations, or performance status limitation will be eligible.

Additionally, those that refuse conventional induction therapy will be eligible.

* Patients must have relatively stable bone marrow function during the week prior to enrollment on the study. White Blood cells (WBC) may be controlled with hydrea. Rapid WBC doubling not responsive to control with hydrea would indicate unstable bone marrow function. Ideally WBC should be < 15 X 10^3 /dl at time of study enrollment.
* Age >18 years
* Karnofsky performance status > or = 60%
* Have acceptable organ function as defined within 28 days of enrollment:

  * Hematologic: hemoglobin > 8 g/dL, and platelets > 20k. (Patients may receive transfusions of either peripheral red blood cells (PRBC) or platelets to achieve these levels)
  * Renal: creatinine < or = 2.0 mg/dL or creatinine clearance > or = 40 ml/min
  * Hepatic: ALT, AST < or = 2.5 x upper limit of normal and total bilirubin < or = 1.5 X ULN
  * Cardiac: left ventricular ejection fraction > 40% (testing required for all patients. For those with prior cardiac history (defined as prior stent or bypass surgery) a stress test within 1 month prior to proceeding with the study will be required. A cardiology consult will be required for those with prior documented cardiac disease or those with any significant EKG/ECHO abnormalities found on screening tests.
* Patients must not have received treatment for their myeloid disorder within 2 weeks of beginning the trial. Treatments include the use of chemotherapy, hematopoietic growth factors, and biologic therapy such as monoclonal antibodies. The exception is the use of hydroxyurea for patients with an elevated WBC. Given the relatively slower expected clinical response with the study drugs, patients may continue to receive hydroxyurea through the first cycle of therapy.
* Must have recovered from clinically significant toxicities from previous therapies.
* Women of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment. In addition, women of childbearing potential must have a negative serum pregnancy test b-hCG within 72 hours prior to receiving the first dose of therapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Treatment History Criteria: Patients who have relapsed after allogeneic stem cell transplantation are eligible.

Exclusion Criteria:

* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test within 72 hours prior to study drug administration to rule out pregnancy.
* Grade 2 or greater peripheral neuropathy within 14 days before enrollment
* Active central nervous system (CNS) disease. Patients with any clinical symptoms of active CNS disease must have LP with negative cytology.
* WBC and Peripheral Blast count uncontrolled with hydroxyurea
* Evidence of QT prolongation with QTc interval greater than 0.5 seconds. QTc calculation from the EKG machine will be used for this assessment.
* Clinical evidence of heart failure or history of uncontrolled hypertension. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patients with untreated positive blood cultures or progressive infections as assessed by radiographic studies
* Patients with prior use of other histone deacetylase inhibitors (excluding valproic acid for seizures with a 30 day wash-out period)
* Known hypersensitivity to Velcade, boron or any of the other agents used in this study
* Patients with a history of deep vein thrombosis/pulmonary embolism (DVT/PE) that has not been adequately treated with systemic anticoagulation or that has been recently diagnosed (within the last 2 months).
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Active HIV or viral hepatitis infection
* Other active and potentially life threatening malignancies excluding localized basal cell or squamous cell skin cancers, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warlick, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study entry is open to patients regardless of gender or ethnic background.
Groups:
- Velcade + Vorinostat in MDS and AML: This is a phase II two stage single arm study combining Velcade on days 1, 4, 8, and 11 plus oral Vorinostat days 1-14 of a 21 days cycle. Treatment will continue for a total of 3 treatment cycles.
  vorinostat : 400 mg orally (po) every day on days 1-14 of a 21 day cycle
  bortezomib : 1.3mg/m^2 via peripheral subcutaneous administration on day 1, 4, 8, 11 of a 21 day cycle
Period: Overall Study
Arm/Group | Velcade + Vorinostat in MDS and AML
Started | 16
Completed | 12
Not Completed | 4
Not completed — Declining performance status | 2
Not completed — Unrelated hip fracture-unable to proceed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Velcade + Vorinostat: This is a phase II two stage single arm study combining Velcade on days 1, 4, 8, and 11 plus oral Vorinostat days 1-14 of a 21 days cycle. Treatment will continue for a total of 3 treatment cycles.
  vorinostat : 400 mg orally (po) every day on days 1-14 of a 21 day cycle
  bortezomib : 1.3mg/m^2 via peripheral subcutaneous administration on day 1, 4, 8, 11 of a 21 day cycle
Arm/Group | Velcade + Vorinostat
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: Years] | 65.5 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients by Best Clinical Response
Description: Assessed by the International Working Group response criteria: Complete Remission - <5% myeloblasts with normal maturation of all cell lines; Partial Remission - bone marrow blasts decreased by > 50% over pre-treatment but still >5%; and Hematologic Improvement - hemoglobin increase by > 1.5g/dl or decreased transfusions by at least 4/8 week period, platelet absolute increase of >30 X 10^9/L for those starting at >20 X 10^9/L . For those < 20 X 10^9 /L at baseline increase by 100%.
Time Frame: At Completion of Course 3 (Day 63)
Population: Evaluable patients are defined as those who completed at least 1 cycle of therapy; 8 had acute myeloid leukemia, 4 had myelodysplastic syndrome.
Measure: Number; unit: Patients
Groups:
- Evaluable Patients: This is a phase II two stage single arm study combining Velcade on days 1, 4, 8, and 11 plus oral Vorinostat days 1-14 of a 21 days cycle. Treatment continued for a total of 3 treatment cycles.
  vorinostat : 400 mg orally (po) every day on days 1-14 of a 21 day cycle
  bortezomib : 1.3mg/m^2 via peripheral subcutaneous administration on day 1, 4, 8, 11 of a 21 day cycle
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 12
Patients
  Complete Remission | 1
  Progressive Disease | 6
  Stable Disease | 5

2. Secondary Outcome: Correlative Laboratory Studies
Description: Analysis of Natural Killer (NK) Cell Activating and Inhibitory Receptor Alterations, NK Cell Receptor Ligand Alterations, HLA Class I Expression on Target Cells (Myeloid Blasts), and NK-mediated Cell Killing
Time Frame: Pre-Study and After 3 Cycles
Population: Natural Killer cell studies were discontinued after the first 3 patients because the results were not helpful, and thus the secondary outcome measures were not completed.
Arm/Group | Velcade + Vorinostat in MDS and AML
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Cell Alterations With Clinical Response
Description: as for outcome 2
Time Frame: Pre-Study and After 3 Cycles
Population: Natural Killer cell studies were discontinued after the first 3 patients because the results were not helpful. So, secondary outcome measures were not completed.
Arm/Group | Velcade + Vorinostat in MDS and AML
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: All patients treated on the trial were included in evaluation of toxicity. Toxicities are defined as non-hematologic given the concurrent impact of AML and MDS on cytopenias.
Arm/Group | Velcade + Vorinostat
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade + Vorinostat (N=16)
Cardiac arrest (Cardiac disorders) | 2 (2)
Ischemia/Elevated Troponin (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade + Vorinostat (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 8 (9)
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (11)
Diplopia (Eye disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (Vascular disorders) | 4 (4)
Elevated ALT/AST/Alkaline Phosphatase (Investigations) | 2 (10)
Elevated creatinine (Investigations) | 4 (10)
Eye pain/blurred vision (Eye disorders) | 2 (2)
Fash rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 9 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (6)
Gingival erythema (Gastrointestinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Hypotension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection, ANC=.03 (Infections and infestations) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Involuntary movements (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemia (Cardiac disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Muscle leg pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea or vomiting (Gastrointestinal disorders) | 9 (17)
Neuropathy (Nervous system disorders) | 4 (5)
Nose bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain upon urination (Renal and urinary disorders) | 1 (1)
Pulmonary infection/pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
QT prolongation (Cardiac disorders) | 6 (9)
Rectal/hemorrhoidal pain (Gastrointestinal disorders) | 1 (1)
Shingles flare (General disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Systolic murmur (Cardiac disorders) | 2 (2)
Tongue blister (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes